CLINICAL TRIAL: NCT07208487
Title: Clinical Study of Pretreatment PET/CT Parameters for Predicting the Efficacy of 125I Seed Implantation in the Treatment of Malignant Tumors
Status: Completed | Type: Observational
Sponsor: Jiangxi Provincial Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2025ky281
Record Dates: First submitted 2025-09-27; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Malignant Tumors
Keywords: 125I seed; Brachytherapy; Malignant tumors; PET/CT; MTV; TLG; SUV; Efficacy prediction
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — CT scans AND PET/CT parameters
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 125I seed implantation treatment group: Inform the patient of relevant precautions and obtain signed informed consent. Upload CT data in DICOM format to the TPS system. Contour the tumor target volume and critical organs layer by layer. Design the needle insertion direction, angle, and depth. Determine the prescribed dose, number of implants, and activity. Obtain the Dose and Volume Histogram (DVH). For patients without prior external beam radiotherapy, the prescribed dose is 120 Gy. For those with prior external beam radiotherapy, the prescribed dose ranges from 80 to 100 Gy, ensuring surrounding critical organs receive doses within safe limits. Position, immobilize, disinfect, and drape the patient according to surgical positioning. After instructing the patient to hold their breath, perform CT scanning for localization. Following local anesthesia, complete particle implantation according to the preoperative plan. After particle implantation, perform another CT scan to verify dose distribution.

SUMMARY:
This study aimed to determine if pre-treatment 18F-FDG PET/CT metabolic parameters could predict the effectiveness of 125I seed implantation for malignant tumors. In a retrospective analysis of 41 patients with 69 lesions, various parameters were measured. The results identified Metabolic Tumor Volume (MTV) as the most significant independent prognostic factor, outperforming other standardized uptake values (SUV) and ratios. A higher MTV was associated with a worse treatment outcome, suggesting it is a valuable predictor for guiding treatment decisions.

DETAILED DESCRIPTION:
Objective The purpose of the research is to assess the role of pretreatment 18F-FDG PET/CT parameters in predicting the efficacy of 125I seed implantation in the treatment of malignant tumors, in order to allow for timely clinical interventions and adjustments in the treatment regimen. Methods A retrospective analysis was made on patients who were treated with 125I seed implantation for malignant tumors and underwent 18F-FDG PET/CT before treatment from November 2019 to November 2023 in our hospital. The clinical data of 41 patients with 69 lesions were collected completely, including age, gender, primary tumor and seed implantation sites. Metabolic parameters including TLG, MTV, SUVmax-bw, SUVmax-bsa, SUVmax-lbm, SUVmean-bw, SUVmean-bsa, SUVmean-lbm, SUVpeak-bw, SUVpeak-bsa, SUVpeak-lbm, TLR, TLMR, TBR and TBMR were measured at pretreatment PET/CT. The patients were followed up at 4 months after the procedure by CT scans. The efficacy of response was evaluated by using the response evaluation criteria in solid tumors (RECIST1.1). Results The area under the curves for TLG and MTV were 0.815 (P<0.001) and 0.804 (P<0.001) respectively. Univariate logistic regression analysis and multivariate logistic regression analysis. The results showed that only the MTV (OR: 6.477, 95%CI: 1.157-36.271, P=0.034) was an independent prognostic factor for the efficacy of 125I seed implantation for malignant tumors. Conclusion In patients with malignant tumors treated with 125I seed implantation, the 18F-FDG PET/CT parameters MTV in the prediction of the efficacy was superior to SUVmax, SUVmean and SUVpeak which normalized by body weight, body surface area and lean body mass, as well as to TLR, TLMR, TBR and TBMR. The 18F-FDG PET/CT parameter MTV was an independent prognostic factor for the efficacy of 125I seed implantation in the treatment of malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

(1) Interval between PET/CT imaging and 125I seed implantation ≤4 weeks; (2)CT follow-up performed 4 months post-125I seed implantation; (3) Primary tumor pathologically or cytologically diagnosed as malignant; (4) Metastatic or recurrent lesions implanted with 125I confirmed by cytological aspiration or imaging

Exclusion Criteria:

(1) Lesions too small or SUVmax < 2.5, rendering them unidentifiable by software for PET/CT parameter measurement; (2) Two 125I seed implantation procedures performed within 6 months for the same lesion; (3) Incomplete clinical or imaging data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with malignant tumors who underwent 125I seed implantation therapy at the Department of Nuclear Medicine, Jiangxi Cancer Hospital between November 2019 and November 2023 and received preoperative 18F-FDG PET/CT scans.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Tumor size | 4 months post-surgery
  Referencing the Response Evaluation Criteria in Solid Tumors (RECIST 1.1), efficacy is categorized as Complete Response (CR), Partial Response (PR), Stable Disease (SD), or Progression Disease (PD). Objective response rate (ORR) was defined as the proportion of lesions achieving CR or PR, while non-ORR was defined as the proportion of lesions achieving SD or PD.

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangxi Cancer Hospital, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Watanabe H, Okada M, Kaji Y, Satouchi M, Sato Y, Yamabe Y, Onaya H, Endo M, Sone M, Arai Y. [New response evaluation criteria in solid tumours-revised RECIST guideline (version 1.1)]. Gan To Kagaku Ryoho. 2009 Dec;36(13):2495-501. Japanese. PMID 20009446